CLINICAL TRIAL: NCT04916171
Title: The Incidence of Endometriosis and or Adenomyosis in Patients Diagnosed With Polycystic Ovary Syndrome, or the Incidence of Polycystic Ovary Syndrome in Patients Diagnosed With Endometriosis and or Adenomyosis
Brief Title: Determination of the Incidence of Endometriosis and or Adenomyosis in Patients Diagnosed With Polycystic Ovary Syndrome, or the Incidence of Polycystic Ovary Syndrome in Patients Diagnosed With Endometriosis and or Adenomyosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Collaborators: Engin Oral (Unknown); Berna Dilbaz (Unknown); Gürkan Bozdag (Unknown); Cem Atabekoğlu (Unknown); Nuray Bozkurt (Unknown); Gokce Anik Ilhan (Unknown); Ali Kolusari (Unknown); Cihan Kaya (Unknown); Banu Yılmaz (Unknown); Engin Yildirim (Unknown); Ahmet Başar Tekin (Unknown); Servet Ozden hacivelioglu (Unknown)
Responsible Party: Principal Investigator, Pınar Yalcin bahat, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: endopcos
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Endometriosis; Polycystic Ovary Syndrome; Adenomyosis
MeSH Terms: conditions — Endometriosis; Polycystic Ovary Syndrome; Adenomyosis | interventions — Incidence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endometriosis and or Adenomyosis in Patients Diagnosed With Polycystic Ovary Syndrome: The diagnosis of endometriosis will be made by the presence of ovarian endometrioma and/or a deep infiltrating endometriosis nodule determined by transvaginal ultrasonography or by palpation of the endometriotic nodule on pelvic examination or surgical confirmation.
  The diagnosis of adenomyosis will be made by transvaginal ultrasonography or surgical confirmation.
  Interventions: Other: incidence
- Polycystic Ovary Syndrome in Patients Diagnosed With Endometriosis and or Adenomyosis: For the diagnosis of polycystic ovary syndrome, Rotterdam Criteria will be used.
  Interventions: Other: incidence

INTERVENTIONS:
Other: incidence — It is aimed to determine the incidence of endometriosis and/or adenomyosis in patients diagnosed with polycystic ovary syndrome, or to determine the incidence of polycystic ovary syndrome in patients diagnosed with endometriosis and/or adenomyosis.

SUMMARY:
The study was designed as a multicenter, prospective cross-sectional cohort study. The research population will consist of patients under the age of 40, diagnosed with endometriosis and/or adenomyosis and polycystic ovary syndrome, who applied to the obstetrics and gynecology outpatient clinics in 13 centers. According to the results of the sample size analysis, it was planned to terminate the study when 1225 patients with polycystic ovary syndrome and 1225 patients with endometriosis and/or adenomyosis were recruited.

DETAILED DESCRIPTION:
For the diagnosis of polycystic ovary syndrome, Rotterdam Criteria will be used. Hyperandrogenism will be determined clinically by Ferriman-Gallwey scoring, and biochemically by serum total testosterone and sex hormone initiating globulin (SHBG). 21-24 and 28-31 of menstruation in patients with ovulatory dysfunction, oligomenorrhea (cycles lasting longer than 38 days). It will be determined by measuring the serum progesterone level between days Polycystic ovarian morphology will be determined by transvaginal ultrasonography (8 mHz probe) by calculating the number of antral follicles and ovarian volume. Serum Anti Mullerian Hormone (AMH) will be requested from patients being investigated for polycystic ovary syndrome.

In order to exclude other conditions during the investigation in patients with suspected polycystic ovary syndrome, serum thyroid stimulating hormone (TSH), prolactin (PRL) and 17-hydroxyprogesterone (17-OHP) levels will be checked in the first 7 days of menstruation.

The diagnosis of endometriosis will be made by the presence of ovarian endometrioma and/or a deep infiltrating endometriosis nodule determined by transvaginal ultrasonography or by palpation of the endometriotic nodule on pelvic examination or surgical confirmation.

The diagnosis of adenomyosis will be made by transvaginal ultrasonography or surgical confirmation.

For polycystic ovary syndrome in patients diagnosed with endometriosis and/or adenomyosis; For endometriosis and/or adenomyosis in patients diagnosed with polycystic ovary syndrome, the above-described diagnostic investigations will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with endometriosis by ultrasound or surgery(after diagnosed)
* Being a newly diagnosed endometriosis patient
* Not using any hormones or additional drugs
* Not having undergone ovarian surgery
* Patients diagnosed with PCOS according to the Rotterdam diagnostic criteria

Exclusion Criteria:

* Previously diagnosed with endometriosis, medically or surgically patients receiving treatment
* Patients who have undergone ovarian surgery

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: The research population will consist of patients under the age of 40, diagnosed with endometriosis and/or adenomyosis and polycystic ovary syndrome, who applied to the obstetrics and gynecology outpatient clinics in 13 centers. According to the results of the sample size analysis, it was planned to terminate the study when 1225 patients with polycystic ovary syndrome and 1225 patients with endometriosis and/or adenomyosis were recruited. For polycystic ovary syndrome in patients diagnosed with endometriosis and/or adenomyosis; For endometriosis and/or adenomyosis in patients diagnosed with polycystic ovary syndrome, the above-described diagnostic investigations will be performed.
Sampling Method: Probability Sample
Enrollment: 2450 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-20 (Estimated)

PRIMARY OUTCOMES:
Demonstration of the co-occurrence of endometriosis, adenomyosis and polycystic ovarian syndrome in women of reproductive age under 40 years of age in our country. | 1 year
  The Co-occurrence rate of endometriosis, adenomyosis and polycystic ovarian syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- Pinar Yalcin Bahat, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided